CLINICAL TRIAL: NCT06320847
Title: Development of Predictive Remote Photoplethysmography Algorithm for Blood Pressure Assessment and Monitoring
Brief Title: Predictive Remote Photoplethysmography Algorithm for Blood Pressure Pressure Assessment and Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Nervotec Pte. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Predictbloodpressure
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Remote Photoplethysmography , Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: rPPG — A pulse oximeter and blood pressure cuff will be applied on the study patient by the study team member (research coordinators). At the same time, vital signs from Nervotec's rPPG technology will be recorded via the laptop and webcam. Synchronous measurement process of heart rate, respiration rate, pulse oximetry, heart rate variability and blood pressure estimates using Nervotec rPPG technology will take place for a duration of 3 minutes.

SUMMARY:
Significant advancements in the field of medical technologies have resulted in the rise of contact-free methods of haemodynamic monitoring. Remote photoplethysmography (rPPG) is a videobased, contactless form of monitoring that operates through a camera-enabled device. This innovation interprets minute variations in skin colour due to blood flow which, when analysed with complex signal processing algorithms, generates vital sign readings. Currently, Nervotec's rPPG technology allows for the collection of rPPG waveforms, which enables the measurement of heart rate, heart rate variability, respiration rate and blood oxygen saturation (SpO2) level through signal processing techniques. The plethysmography signals can be used to estimate blood pressure through the creation and training of a predictive model. By examining and extracting key features of a continuous PPG waveform by training an artificial neural network, correlations between these features and BP can be studied.

DETAILED DESCRIPTION:
This is a prospective, feasibility study.Background literature has shown that plethysmography (PPG) signals can be used to estimate blood pressure through the creation and training of a predictive model. By examining and extracting key features of a continuous PPG waveform by training an artificial neural network, correlations between these features and blood pressure can be studied.

Nervotec, a digital health and AI company , has successfully used rPPG technology to allow for collection of rPPG waveforms, which enables the measurement of heart rate (HR), heart rate variability (HRV), respiration rate (RR) and blood oxygen saturation (SpO2) level through signal processing techniques. They have incorporated rPPG technology into a mobile application using smartphone cameras for scanning an individual's face. However, this is yet to be established for blood pressure. We aim to perform a prospective study to evaluate the feasibility and accuracy of obtaining blood pressure measurements through rPPG.

Hypothesis: Remote photoplethysmography can be used to determine blood pressure and this algorithm can develop into a customised smartphone based application.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years old
* Ability to provide informed consent
* Any surgery except head and neck surgeries

Exclusion Criteria:

* Age ≤ 21 years old
* Inability to provide informed consent
* Patients going for head and neck surgery

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To determine the correlation between remote photoplethysmography (rPPG) and blood pressure variations. | 1 year
To develop a predictive model in using rPPG for determination of blood pressure. | 1 year
To validate this predictive model by comparing blood pressure readings obtained using rPPG with standard procedures such as contact sensors and automated oscillometry. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore